CLINICAL TRIAL: NCT02262832
Title: Compassionate Use of Metreleptin in Previously-Treated Patients With Generalized Lipodystrophy
Brief Title: Compassionate Use of Metreleptin in Previously Treated People With Generalized Lipodystrophy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150003; 15-DK-0003
Record Dates: First submitted 2014-10-10; First posted 2014-10-13 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-11-20

CONDITIONS: Lipodystrophy; Diabetes; Hyperlipidemia
Keywords: Diabetes; Leptin; Lipodystrophy; Hypertriglyceridemia
MeSH Terms: conditions — Lipodystrophy; Diabetes Mellitus; Hyperlipidemias; Hypertriglyceridemia | interventions — metreleptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Leptin study drug (Other): Administration of study drug SQ BID
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — administered subcutaneously 1-2 times/day

SUMMARY:
Background:

- Generalized lipodystrophy can cause high blood fat levels and resistance to insulin. This can lead to health problems including diabetes. Researchers have found that the drug metreleptin improves health in people with this disease.

Objective:

- To test the safety and effectiveness of metreleptin.

Eligibility:

* People ages 6 months and older with generalized lipodystrophy who:
* have received metreleptin through NIH studies AND
* cannot get it through approved or compassionate use mechanisms in their home country.

Design:

* Participants will come to NIH approximately every 6 months during year one, then every 1 2 years. Financial assistance may be available for travel within the U.S.
* At visits, participants will get a supply of metreleptin to take home for daily injections. They will have:
* plastic catheter placed in an arm vein.
* blood tests, urine collection, and physical exam.
* oral glucose tolerance test, drinking a sweet liquid.
* ultrasound of the heart, liver, uterus, and ovaries. A gel and a probe are placed on the skin and pictures are taken of the organs.
* echocardiogram, which takes pictures of the heart with sound waves.
* Resting Metabolic Rate taken. A plastic hood is worn over the head while the oxygen they breathe is measured.
* Participants will have up to 3 DEXA scan x-rays per year.
* Participants may have:
* annual bone x-rays.
* liver biopsies every few years. A needle will be inserted into the liver to obtain a small piece. Participants will sign a separate consent for this.
* Participants must be seen regularly by their local doctors and have blood tests at least every 3 6 months at home.

DETAILED DESCRIPTION:
Leptin is an adipocyte-derived hormone that can be thought of as a signal from adipose tissue to the rest of the body conveying information about long-term nutritional status. Patients with the very rare condition of generalized lipodystrophy have leptin deficiency secondary to lack of adipose tissue. The combination of leptin deficiency and ectopic lipid deposition in patients with lipodystrophy leads to metabolic complications including severe insulin resistance and diabetes, hypertriglyceridemia, nonalcoholic steatohepatitis, and polycystic ovarian syndrome. Between 2000 and 2014, the NIDDK IRP conducted an open-label clinical trial of the recombinant human leptin analog, metreleptin, in patients with generalized and partial forms of lipodystrophy. This study showed that metreleptin ameliorates metabolic and endocrine abnormalities in lipodystrophy, including reducing food intake, improving insulin resistance and diabetes, reducing ectopic lipid, and normalizing reproduction. Based on these data, metreleptin was approved by the FDA in February, 2014, for patients with generalized, but not partial, lipodystrophy.

Currently, metreleptin is not available as an approved drug outside the US and Japan, and it is available on a compassionate use basis only in a few additional countries. The purpose of this study is twofold:

1. To provide access to metreleptin to patients with generalized lipodystrophy, including those who have previously received metreleptin through NIH studies (protocols 02-DK-0022 and 13-DK- 0057) AND/OR who cannot obtain metreleptin through approved or compassionate use mechanisms in their home country
2. To continue to collect data on the long-term efficacy of metreleptin in ameliorating the metabolic complications of generalized lipodystrophy.

Metreleptin will be given at doses of less than or equal to 0.24 mg/kg/day, adjusted based on body weight and metabolic control. Patients will be seen approximately once per year at NIH for evaluation, and potentially less frequently for those who are medically stable and have difficulty traveling to the US. Laboratory evaluation will be obtained more frequently by the patient s home providers as clinically indicated. The primary outcomes of the study are improvements in serum triglycerides and hemoglobin A1c levels. Secondary outcomes include measures of steatohepatitis and ectopic lipid, body composition, bone mineral density and bone mineral metabolism, and pituitary and reproductive function.

Metreleptin is supplied by Chiesi USA, Inc.. Neither the NIH nor Chiesi USA, Inc. can guarantee that leptin will be available for these patients indefinitely and/or after the study ends.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 6 months.
  2. Generalized lipodystrophy (either congenital or acquired).
  3. Those who cannot obtain metreleptin through approved or compassionate use mechanisms in their home country.

EXCLUSION CRITERIA:

1. Availability of metreleptin to the patient either as an approved drug, or through local compassionate use or expanded access programs.
2. Known HIV infection or HIV-associated lipodystrophy.
3. Any medical condition or medication that will increase risk to the subject.
4. Current alcohol or substance abuse.
5. Subjects who have a known hypersensitivity to E. coli derived proteins (as leptin is derived from such proteins).

Ages: 6 Months to 98 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Serum triglycerides | every 6-12 months
  Improvements in lab value.
Serum hemoglobin A1C | every 6-12 months
  Improvements in lab value.

SECONDARY OUTCOMES:
Steatohepatosis | every 12 months
  stable or improvements
Pituitary & Reproductive Function | every 6-12 months
  stable or improvements
Ectopic lipid & body composition | every 12 months
  stable or improvements
Bone mineral density & metabolism | every 12 months
  stable or improvements

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- [Background] Malandrino N, Reynolds JC, Brychta RJ, Chen KY, Auh S, Gharib AM, Startzell M, Cochran EK, Brown RJ. Visceral fat does not contribute to metabolic disease in lipodystrophy. Obes Sci Pract. 2019 Jan 24;5(1):75-82. doi: 10.1002/osp4.319. eCollection 2019 Feb. PMID 30847226
- [Background] Meral R, Ryan BJ, Malandrino N, Jalal A, Neidert AH, Muniyappa R, Akinci B, Horowitz JF, Brown RJ, Oral EA. "Fat Shadows" From DXA for the Qualitative Assessment of Lipodystrophy: When a Picture Is Worth a Thousand Numbers. Diabetes Care. 2018 Oct;41(10):2255-2258. doi: 10.2337/dc18-0978. PMID 30237235
- [Derived] Brown RJ, Meehan CA, Cochran E, Rother KI, Kleiner DE, Walter M, Gorden P. Effects of Metreleptin in Pediatric Patients With Lipodystrophy. J Clin Endocrinol Metab. 2017 May 1;102(5):1511-1519. doi: 10.1210/jc.2016-3628. PMID 28324110
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-DK-0003.html